CLINICAL TRIAL: NCT00477152
Title: INcreased Flow Utilizing Subcutaneously-Enabled Pediatric Rehydration (INFUSE-Pediatric Rehydration Study): Phase IV Study of Subcutaneous Rehydration With Recombinant Human Hyaluronidase (HYLENEX) for Infants and Children
Brief Title: Study of Subcutaneous Rehydration With Recombinant Human Hyaluronidase for Infants and Children
Acronym: INFUSE-PR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Halozyme Therapeutics (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1838-003
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2011-11-23 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Dehydration
Keywords: dehydration; fluid therapy; pediatrics; emergency medicine; hyaluronoglucosaminidase; hyaluronidase; hypodermoclysis; clysis; subcutaneous hydration; subcutaneous rehydration; hyaluronan; rHuPH20
MeSH Terms: conditions — Dehydration | interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HYLENEX-augmented subcutaneous (SC ) rehydration (Experimental): Single 150 U subcutaneous (SC) HYLENEX dose administered immediately prior to start of SC infusion of rehydration fluid. Additional 150 U HYLENEX dose to be administered prior to any additional fluid infusion beyond 24 hours.
  Interventions: Drug: hyaluronidase (human recombinant)/rehydration fluid

INTERVENTIONS:
Drug: hyaluronidase (human recombinant)/rehydration fluid — Single 150 U subcutaneous (SC) HYLENEX dose administered immediately prior to start of SC infusion of rehydration fluid. Additional 150 U HYLENEX dose to be administered prior to any additional fluid infusion beyond 24 hours.
  Other Names: HYLENEX recombinant

SUMMARY:
The aim of the study is to evaluate the safety, effectiveness and ease of use of subcutaneous (SC) rehydration using HYLENEX-augmented SC infusion of fluids and electrolytes for the rehydration of pediatric patients with mild to moderate dehydration.

DETAILED DESCRIPTION:
Pediatric patients (2 months to 10 years of age), presenting to the emergency department (ED) with mild to moderate dehydration and requiring parenteral rehydration, were treated with HYLENEX-augmented subcutaneous (SC) rehydration. An initial volume of 20 mL/kg of isotonic fluid was to be administered by continuous SC infusion over the first hour, and additional SC rehydration could be continued as clinically indicated. The preferred anatomic site for the SC infusion was the anterior thigh, unless there was an overriding preference for an alternate site.

The duration of HYLENEX-augmented SC rehydration was to be a minimum of 1 hour and a maximum of 72 hours. The investigator or designee performed a clinical assessment of the subject's hydration status at baseline and at the end of SC infusion or at discharge from the ED. Other assessments of effectiveness and safety were made directly during the rehydration period and ED stay, and by telephone on Days 3 and 7 after discharge from the ED.

ELIGIBILITY:
Inclusion Criteria:

* Child, 2 months to 10 years of age
* Body weight less than 42 kg
* Presenting at emergency department with mild to moderate dehydration (Gorelick dehydration classification: presence of 1 to 6 [of possible 10] moderate or severe signs and symptoms) requiring parenteral rehydration

Exclusion Criteria:

* In shock or life-threatening situation (other than dehydration)
* Severe dehydration
* Requires intravenous (IV) therapy for another indication
* Indwelling IV catheter (excepting one intended strictly for clinical laboratory sample collection)
* Already received rehydration therapy IV within prior 48 hours or substantial oral fluid immediately before enrollment
* Condition precluding subcutaneous injection or infusion site evaluation in anterior thigh or other elected infusion site
* Reason for hospital admission or extended emergency department stay other than dehydration
* Known hypersensitivity to hyaluronidase or another ingredient in HYLENEX
* Hyponatremia or hypernatremia
* Hypokalemia
* Medical condition likely to interfere with ability to fully complete study or have protocol-specified assessments
* Medical history, screening examination finding or historical clinical laboratory result precluding safe participation in study or which might adversely effect interpretation of study results
* Participated in study of any investigational drug or device within 30 days prior to this study

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George E Harb, MD, Study Director — Baxter Healthcare Corporation

REFERENCES:
- [Background] Gorelick MH, Shaw KN, Murphy KO. Validity and reliability of clinical signs in the diagnosis of dehydration in children. Pediatrics. 1997 May;99(5):E6. doi: 10.1542/peds.99.5.e6. PMID 9113963
- [Result] Allen CH, Etzwiler LS, Miller MK, Maher G, Mace S, Hostetler MA, Smith SR, Reinhardt N, Hahn B, Harb G; INcreased Flow Utilizing Subcutaneously-Enabled Pediatric Rehydration Study Collaborative Research Group. Recombinant human hyaluronidase-enabled subcutaneous pediatric rehydration. Pediatrics. 2009 Nov;124(5):e858-67. doi: 10.1542/peds.2008-3588. Epub 2009 Oct 5. PMID 19805455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited in emergency department after presenting with signs of mild to moderate dehydration
Groups:
- HYLENEX-augmented Subcutaneous (SC) Rehydration: Single 150 U subcutaneous (SC) HYLENEX dose administered immediately prior to start of SC infusion of rehydration fluid. Additional 150 U HYLENEX dose to be administered prior to any additional fluid infusion beyond 24 hours.
Period: Overall Study
Arm/Group | HYLENEX-augmented Subcutaneous (SC) Rehydration
Started | 52 (One patient withdrawn prior to treatment, so not included in analyses.)
Completed | 49 (Two patients treated, but assessments incomplete. All available data included in analyses for these.)
Not Completed | 3
Not completed — Parent withdrew consent | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | HYLENEX-augmented Subcutaneous (SC) Rehydration
Number analyzed (Participants) | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 1.91 (1.949)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 51
Age Categorical [Number; unit: participants]
  >= 2 months to < 3 years | 43
  >= 3 years to <= 10 years | 8
Gorelick Dehydration Score [Mean (Standard Deviation); unit: Number of moderate/severe symptoms] — Score indicates the number of moderate-to-severe signs/symptoms of dehydration, based on assessment of each of the following ten patient parameters: general condition, quality of radial pulse, quality of respiration, skin elasticity, eyes, tears, mucous membranes, urine output, heart rate and fingertip capillary refill time. Minimum score = 0; maximum score = 10. (Note: study inclusion criterion required a baseline score of 1 to 6.)
  Number of moderate/severe symptoms | 3.5 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: HYLENEX-facilitated Subcutaneous (SC) Rehydration Success
Description: Successfully rehydrated (as medically judged by treating physician) without rescue therapy (ie, without receiving fluids via an alternate route), and discharged to home
Time Frame: At emergency department discharge (mean time to discharge = 7.03 ± 7.57 hr)
Population: ITT (all treated patients)
Measure: Number; unit: participants
Arm/Group | HYLENEX-augmented Subcutaneous (SC) Rehydration
Number analyzed (Participants) | 51
participants | 43

2. Primary Outcome: Modified HYLENEX-facilitated Subcutaneous (SC) Rehydration Success
Description: Successfully rehydrated (as medically judged by treating physician) without rescue therapy (ie, without receiving fluids via an alternate route), regardless of emergency department discharge destination
Time Frame: At emergency department discharge (mean time to discharge = 7.03 ± 7.57 hr)
Population: ITT (all treated patients)
Measure: Number; unit: participants
Arm/Group | HYLENEX-augmented Subcutaneous (SC) Rehydration
Number analyzed (Participants) | 51
participants | 48

3. Secondary Outcome: Number of Attempts Needed to Successfully Place Subcutaneous (SC) Catheter
Time Frame: At end of placement of SC catheter
Population: ITT (all treated patients)
Measure: Number; unit: participants
Arm/Group | HYLENEX-augmented Subcutaneous (SC) Rehydration
Number analyzed (Participants) | 51
participants
  1 attempt | 46
  2 attempts | 5

4. Secondary Outcome: Post-treatment Gorelick Dehydration Score
Description: Score indicates the number of moderate-to-severe signs/symptoms of dehydration, based on assessment of each of the following 10 patient parameters: general condition, quality of radial pulse, quality of respiration, skin elasticity, eyes, tears, mucous membranes, urine output, heart rate and fingertip capillary refill time. Minimum score = 0; maximum score = 10.
Time Frame: At baseline and at either the end of subcutaneous infusion (mean duration = 5.73 ± 9.15 hr) or emergency department discharge (mean time to discharge = 7.03 ± 7.57 hr)
Population: ITT (all treated patients)
Measure: Mean (Standard Deviation); unit: No. moderate/severe symptoms (max = 10)
Arm/Group | HYLENEX-augmented Subcutaneous (SC) Rehydration
Number analyzed (Participants) | 51
No. moderate/severe symptoms (max = 10)
  Actual Score | 0.5 (0.9)
  Change from Baseline | -3.0 (1.2)

ADVERSE EVENTS:
Arm/Group | HYLENEX-augmented Subcutaneous (SC) Rehydration
Serious Adverse Events (participants affected / at risk) | 1/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HYLENEX-augmented Subcutaneous (SC) Rehydration (N=51)
Infusion site cellulitis (Infections and infestations) | 1 (1) — Unrelated to HYLENEX
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HYLENEX-augmented Subcutaneous (SC) Rehydration (N=51)
Infusion site erythema (General disorders) | 44
Infusion site haemorrhage (General disorders) | 2
Infusion site pain (General disorders) | 46
Infusion site rash (General disorders) | 2
Infusion site swelling (General disorders) | 51
Pyrexia (General disorders) | 2
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs vary per individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (eg, for confidential information) up to 90 days prior to submission or communication. Baxter may request an additional delay of up to 60 days (eg, to allow for intellectual property protection).